CLINICAL TRIAL: NCT03276637
Title: The MilSeq Project: Enabling Personalized Medicine Through Exome Sequencing in the U.S. Air Force
Brief Title: Enabling Personalized Medicine Through Exome Sequencing in the U.S. Air Force
Acronym: MilSeq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Professor of Medicine, Division of Genetics, Department of Medicine, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: The MilSeq Project
Record Dates: First submitted 2017-08-31; First posted 2017-09-08 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Healthy Adults; Genetic Predisposition to Disease
Keywords: Whole Genome Sequencing; Whole Exome Sequencing; Military; Air Force; Disease Susceptibility; Genetic Predisposition to Disease; Disease Attributes; Pathologic Processes
MeSH Terms: conditions — Genetic Predisposition to Disease; Disease Susceptibility; Disease Attributes; Pathologic Processes | interventions — Exome Sequencing

STUDY DESIGN:
Intervention Model Description: Whole exome sequencing (WES) will be performed on 75 ostensibly healthy, active-duty Airmen (patient-participants) who receive medical care in military Primary Care, Internal Medicine and/or Family Practice settings who in their baseline survey expressed interest in receiving WES. Military healthcare providers who have received brief genomics training will return results to the patient-participants and the WES reports will be permanently integrated into their electronic medical record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Active-Duty Airmen Cohort (Experimental): Whole exome sequencing (WES) will be performed on 75 ostensibly healthy, active-duty Airmen (patient-participants) who receive medical care in military Primary Care, Internal Medicine and/or Family Practice settings who in their baseline survey expressed interest in receiving WES. Military healthcare providers who have received brief genomics training will return results to the patient-participants and the WES reports will be permanently integrated into their electronic medical record.
  Interventions: Genetic: Whole exome sequencing
- Healthcare Provider Cohort (No Intervention): The Healthcare providers who provide medical care in military Primary Care, Internal Medicine and/or Family Practice settings and enroll participants. Military healthcare providers have received a brief genomics training and will return results to the patient-participants

INTERVENTIONS:
Genetic: Whole exome sequencing — Whole exome sequencing at 125x coverage (i.e., at least 125 sequencing reads covering each position within the exome region of interest) performed at the Laboratory of Molecular Medicine's Clinical Laboratory Improvement Amendments (CLIA) certified laboratory on 75 enrolled individuals
  Arms: Healthy Active-Duty Airmen Cohort

SUMMARY:
The MilSeq Project is a nonrandomized, prospective pilot study of whole exome sequencing (WES) in the U.S. Air Force. The purpose of this study is to explore the implementation of WES into clinical medical care in the military health system.

DETAILED DESCRIPTION:
The objective of this effort is to investigate: (a) military healthcare providers' (HCPs') genomic knowledge before and after receiving a genomic educational primer and after disclosing whole exome sequencing (WES) results to begin to assess the genomic educational needs of military HCPs; (b) active-duty Airmen's knowledge and perceptions of genomic sequencing (GS); (c) reasons why active-duty Airmen choose to participate, or not to participate, in research involving GS; (d) how WES study participants, including HCPs and sequenced active-duty Airmen (patient-participants), respond to and use WES results; (e) the collection of medical, behavioral, and healthcare utilization outcomes related to the clinical integration of WES in the military; (f) how return of WES results and integration into the Electronic Medical Record (EMR) do or do not impact perceptions of mission readiness and duty assignments. Given the lack of prior research in this area in the Air Force and the broad number of topics of interest, the aims of the study are predominantly exploratory and results may be hypothesis generating.

The MilSeq Project will be conducted in two sequential phases. Phase I of the study will recruit, consent, and enroll approximately 75 ostensibly healthy active-duty Airmen who receive medical care in military Primary Care, Internal Medicine, and/or Family Practice settings to take a baseline survey. This survey will be administered to explore active-duty Airmen's perceptions of and preferences for GS, identify motivations and barriers to active-duty Airmen participating in a WES study, and assess interest in taking part in the WES study.

Phase II of the study will recruit, consent, and enroll 75 ostensibly healthy active-duty Airmen who receive medical care in military Primary Care, Internal Medicine and/or Family Practice settings who in their baseline survey expressed interest in receiving WES through a research study. WES will be performed on each enrolled patient-participant. The result will be disclosed by an HCP-participant and permanently integrated into the patient-participant's EMR. Phase II will also recruit 10-20 military Primary Care, Internal Medicine, and/or Family Practice HCPs and consent them to participate in the study. The HCPs will receive an educational primer in genomics and will disclose WES results to Airmen participants.

There are a number of potential benefits and challenges to incorporating genomic medicine into the military, some that are relevant to the broader civilian community, but some that are unique to this population. Some of these challenges include: (a) how GS may or may not affect the perception of fitness for duty; (b) how genomic discrimination may or may not occur in the military setting; (c) how to best deal with unanticipated findings; and (d) how genomic results can be practically integrated into a military setting. In this pilot study, these potential opportunities and challenges will be explored, which will provide a basis for future study and begin to inform decisions regarding clinical care of active-duty service members.

ELIGIBILITY:
Patient-Participant Inclusion Criteria:

* 18 years or older
* An active Air Force Airman
* Fluent in English
* Seen or eligible to be seen by a provider at Wilford Hall Ambulatory Surgical Center at Joint Base San Antonio (JBSA) Lackland Air Force Base

Healthcare Provider-Participant Inclusion Criterion

* An active or Department of Defense civilian Primary Care, Internal Medicine, or Family Practice Healthcare Provider (Physician, Physician Assistant, or Nurse Practitioner) or resident practicing at Wilford Hall Ambulatory Surgical Center at JBSA Lackland Air Force Base

Patient-Participant Exclusion Criteria:

* Those who do not meet the above inclusion criteria
* Those with clinically concerning scores on anxiety and distress scales in baseline survey
* Trainees (basic military training or tech school)
* Airmen with an active change of duty station order or deployment order and expected to leave San Antonio in 6 months or less
* Airmen expected to be discharged from the Air Force in 6 months or less

Healthcare Provider-Participant Exclusion Criteria:

* Providers who do not meet the above inclusion criteria
* Providers with an active change of duty station order or deployment order and expected to leave San Antonio in 6 months or less
* Providers expected to be discharged from the Air Force in 6 months or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-06-22 (Actual); Study Completion 2020-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas
  - Joint Base San Antonio Lackland Air Force Base - 59th Medical Wing, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McMorrow D. The $100 genome: implications for the DoD. Technical Report. McLean, Virginia: The MITRE Corporation; 2010.
- [Background] De Castro M, Biesecker LG, Turner C, Brenner R, Witkop C, Mehlman M, Bradburne C, Green RC. Genomic medicine in the military. NPJ Genom Med. 2016 Jan 13;1:15008. doi: 10.1038/npjgenmed.2015.8. eCollection 2016. PMID 29263806
- [Background] Collins FS, Guttmacher AE. Genetics moves into the medical mainstream. JAMA. 2001 Nov 14;286(18):2322-4. doi: 10.1001/jama.286.18.2322. No abstract available. PMID 11710899
- [Background] Collins FS, Green ED, Guttmacher AE, Guyer MS; US National Human Genome Research Institute. A vision for the future of genomics research. Nature. 2003 Apr 24;422(6934):835-47. doi: 10.1038/nature01626. Epub 2003 Apr 14. No abstract available. PMID 12695777
- [Background] McCarthy JJ, McLeod HL, Ginsburg GS. Genomic medicine: a decade of successes, challenges, and opportunities. Sci Transl Med. 2013 Jun 12;5(189):189sr4. doi: 10.1126/scitranslmed.3005785. PMID 23761042
- [Background] Green RC, Rehm HL, Kohane IS. Clinical genome sequencing. In: Ginsburg GS, Willard HF, eds. Genomic and Personalized Medicine. 2nd ed. San Diego: Academic Press; 2013:102-22.
- [Background] Christensen KD, Vassy JL, Jamal L, Lehmann LS, Slashinski MJ, Perry DL, Robinson JO, Blumenthal-Barby J, Feuerman LZ, Murray MF, Green RC, McGuire AL; MedSeq Project Team. Are physicians prepared for whole genome sequencing? a qualitative analysis. Clin Genet. 2016 Feb;89(2):228-34. doi: 10.1111/cge.12626. Epub 2015 Jul 7. PMID 26080898
- [Background] Vassy JL, Christensen KD, Slashinski MJ, Lautenbach DM, Raghavan S, Robinson JO, Blumenthal-Barby J, Feuerman LZ, Lehmann LS, Murray MF, Green RC, McGuire AL. 'Someday it will be the norm': physician perspectives on the utility of genome sequencing for patient care in the MedSeq Project. Per Med. 2015;12(1):23-32. doi: 10.2217/pme.14.68. PMID 25642274
- [Background] Vassy JL, Lautenbach DM, McLaughlin HM, Kong SW, Christensen KD, Krier J, Kohane IS, Feuerman LZ, Blumenthal-Barby J, Roberts JS, Lehmann LS, Ho CY, Ubel PA, MacRae CA, Seidman CE, Murray MF, McGuire AL, Rehm HL, Green RC; MedSeq Project. The MedSeq Project: a randomized trial of integrating whole genome sequencing into clinical medicine. Trials. 2014 Mar 20;15:85. doi: 10.1186/1745-6215-15-85. PMID 24645908
- [Background] Johnston JJ, Lewis KL, Ng D, Singh LN, Wynter J, Brewer C, Brooks BP, Brownell I, Candotti F, Gonsalves SG, Hart SP, Kong HH, Rother KI, Sokolic R, Solomon BD, Zein WM, Cooper DN, Stenson PD, Mullikin JC, Biesecker LG. Individualized iterative phenotyping for genome-wide analysis of loss-of-function mutations. Am J Hum Genet. 2015 Jun 4;96(6):913-25. doi: 10.1016/j.ajhg.2015.04.013. PMID 26046366
- [Background] Green RC, Lautenbach D, McGuire AL. GINA, genetic discrimination, and genomic medicine. N Engl J Med. 2015 Jan 29;372(5):397-9. doi: 10.1056/NEJMp1404776. No abstract available. PMID 25629736
- [Background] Robinson JO, Carroll TM, Feuerman LZ, Perry DL, Hoffman-Andrews L, Walsh RC, Christensen KD, Green RC, McGuire AL; MedSeq Project Team. Participants and Study Decliners' Perspectives About the Risks of Participating in a Clinical Trial of Whole Genome Sequencing. J Empir Res Hum Res Ethics. 2016 Feb;11(1):21-30. doi: 10.1177/1556264615624078. Epub 2016 Feb 28. PMID 26928896
- [Background] Vassy JL, McLaughlin HM, MacRae CA, Seidman CE, Lautenbach D, Krier JB, Lane WJ, Kohane IS, Murray MF, McGuire AL, Rehm HL, Green RC. A one-page summary report of genome sequencing for the healthy adult. Public Health Genomics. 2015;18(2):123-9. doi: 10.1159/000370102. Epub 2015 Jan 21. PMID 25612602
- [Background] Krier J, McLaughlin HM, Lane WJ, et al. The return of pharmacogenomic variants in the MedSeq Project: reporting approach and physician response. Annual Meeting of the American Society of Human Genetics. Boston, MA2013
- [Background] Lane WJ, Westhoff CM, Uy JM, Aguad M, Smeland-Wagman R, Kaufman RM, Rehm HL, Green RC, Silberstein LE; MedSeq Project. Comprehensive red blood cell and platelet antigen prediction from whole genome sequencing: proof of principle. Transfusion. 2016 Mar;56(3):743-54. doi: 10.1111/trf.13416. Epub 2015 Dec 3. PMID 26634332
- [Background] Giovanni MA, Krier J, Vassy JL, Lautenbach DM, Green RC, Murray MF. A brief curriculum for physician orientation to clinical whole genome sequencing. American Society of Human Genetics Annual Meeting. Boston, MA2013.
- [Background] Krier JB, Blout CB, D L, et al. Communication and management of genomic sequencing results by non-geneticist physicians. American Society of Human Genetics; 2015; Baltimore, MD.
- [Background] Green RC, Goddard KAB, Jarvik GP, Amendola LM, Appelbaum PS, Berg JS, Bernhardt BA, Biesecker LG, Biswas S, Blout CL, Bowling KM, Brothers KB, Burke W, Caga-Anan CF, Chinnaiyan AM, Chung WK, Clayton EW, Cooper GM, East K, Evans JP, Fullerton SM, Garraway LA, Garrett JR, Gray SW, Henderson GE, Hindorff LA, Holm IA, Lewis MH, Hutter CM, Janne PA, Joffe S, Kaufman D, Knoppers BM, Koenig BA, Krantz ID, Manolio TA, McCullough L, McEwen J, McGuire A, Muzny D, Myers RM, Nickerson DA, Ou J, Parsons DW, Petersen GM, Plon SE, Rehm HL, Roberts JS, Robinson D, Salama JS, Scollon S, Sharp RR, Shirts B, Spinner NB, Tabor HK, Tarczy-Hornoch P, Veenstra DL, Wagle N, Weck K, Wilfond BS, Wilhelmsen K, Wolf SM, Wynn J, Yu JH; CSER Consortium. Clinical Sequencing Exploratory Research Consortium: Accelerating Evidence-Based Practice of Genomic Medicine. Am J Hum Genet. 2016 Jun 2;98(6):1051-1066. doi: 10.1016/j.ajhg.2016.04.011. Epub 2016 May 12. PMID 27181682
- [Background] Berg JS, Agrawal PB, Bailey DB Jr, Beggs AH, Brenner SE, Brower AM, Cakici JA, Ceyhan-Birsoy O, Chan K, Chen F, Currier RJ, Dukhovny D, Green RC, Harris-Wai J, Holm IA, Iglesias B, Joseph G, Kingsmore SF, Koenig BA, Kwok PY, Lantos J, Leeder SJ, Lewis MA, McGuire AL, Milko LV, Mooney SD, Parad RB, Pereira S, Petrikin J, Powell BC, Powell CM, Puck JM, Rehm HL, Risch N, Roche M, Shieh JT, Veeraraghavan N, Watson MS, Willig L, Yu TW, Urv T, Wise AL. Newborn Sequencing in Genomic Medicine and Public Health. Pediatrics. 2017 Feb;139(2):e20162252. doi: 10.1542/peds.2016-2252. Epub 2017 Jan 17. PMID 28096516
- [Background] Kaphingst KA, Facio FM, Cheng MR, Brooks S, Eidem H, Linn A, Biesecker BB, Biesecker LG. Effects of informed consent for individual genome sequencing on relevant knowledge. Clin Genet. 2012 Nov;82(5):408-15. doi: 10.1111/j.1399-0004.2012.01909.x. Epub 2012 Aug 7. PMID 22694298
- [Background] Bowling BV, Acra EE, Wang L, Myers MF, Dean GE, Markle GC, Moskalik CL, Huether CA. Development and evaluation of a genetics literacy assessment instrument for undergraduates. Genetics. 2008 Jan;178(1):15-22. doi: 10.1534/genetics.107.079533. PMID 18202354
- [Background] Gray SW, Hicks-Courant K, Cronin A, Rollins BJ, Weeks JC. Physicians' attitudes about multiplex tumor genomic testing. J Clin Oncol. 2014 May 1;32(13):1317-23. doi: 10.1200/JCO.2013.52.4298. Epub 2014 Mar 24. PMID 24663044
- [Background] Selim AJ, Rogers W, Qian SX, Brazier J, Kazis LE. A preference-based measure of health: the VR-6D derived from the veterans RAND 12-Item Health Survey. Qual Life Res. 2011 Oct;20(8):1337-47. doi: 10.1007/s11136-011-9866-y. Epub 2011 Feb 19. PMID 21336657

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Active-Duty Airmen Cohort | Healthcare Provider Cohort
Started (Completed baseline survey) | 93 | 12
Airmen Pre Survey | 93 | 0
Underwent Sequencing | 75 | 0
Airmen Post Survey | 69 | 0
HCP Pre Survey | 0 | 12
HCP Post Survey | 0 | 12
Completed (Completed follow-up survey) | 69 | 12
Not Completed | 24 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Active-Duty Airmen Cohort: Whole exome sequencing (WES) will be performed on 75 ostensibly healthy, active-duty Airmen (patient-participants) who receive medical care in military Primary Care, Internal Medicine and/or Family Practice settings who in their baseline survey expressed interest in receiving WES. Military healthcare providers who have received brief genomics training will return results to the patient-participants and the WES reports will be permanently integrated into their electronic medical record.
  Whole exome sequencing: Whole exome sequencing at 125x coverage (i.e., at least 125 sequencing reads covering each position within the exome region of interest) performed at the Laboratory of Molecular Medicine's CLIA certified laboratory on 75 enrolled individuals
- Total: Total of all reporting groups
Arm/Group | Healthy Active-Duty Airmen Cohort | Healthcare Provider Cohort | Total
Number analyzed (Participants) | 93 | 12 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 12 | 105
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.75 (8.3) | 39 (9.25) | 34.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 4 | 49
  Male | 48 | 8 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic or Lation | 17 | 0 | 17
  Race/Ethnicity: Non-Hispanic White | 61 | 6 | 67
  Race/Ethnicity: Non-Hispanic Other | 13 | 6 | 19
  Race/Ethnicity: Prefer Not to Answer | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 93 | 12 | 105

OUTCOME MEASURES:

1. Primary Outcome: Active-duty Airmen's Perceptions About Military Use of Genomic Information to Make Career Decisions
Description: Assessed using a novel measure of perceptions about use of genetic information for military career duty assignment decisions on a 1-5 scale, where higher scores indicate more positive attitudes.
Time Frame: Baseline and 6 weeks post disclosure of genomic sequencing results (approx. 43 weeks after baseline)
Population: 69 participants completed follow-up survey
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthy Active-Duty Airmen Cohort: Ostensibly healthy, active-duty Airmen who receive medical care in military Primary Care, Internal Medicine and/or Family Practice settings who in their baseline survey expressed interest in receiving exome sequencing (ES) undergo ES and have the results returned to them.
Arm/Group | Healthy Active-Duty Airmen Cohort
Number analyzed (Participants) | 75
score on a scale
  Baseline | 2.62 (0.75)
  6-weeks post-disclosure | 2.66 (0.91)

2. Primary Outcome: Genomic Sequencing Findings
Description: Analysis of whole exome sequencing results identified the number of participants with genomic findings, including monogenic disease risk, carrier status, and risk allele presence.
Time Frame: Results disclosure (within 1 month of sequencing completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Active-Duty Airmen Cohort
Number analyzed (Participants) | 75
Participants
  Monogenic disease findings: Present | 11
  Monogenic disease findings: Not Present | 64
  Carrier status findings: Present | 65
  Carrier status findings: Not Present | 10
  Risk Allele findings: Present | 37
  Risk Allele findings: Not Present | 38

3. Primary Outcome: Active-duty Airmen Reported Health Care Utilization Related to Study Results
Description: Participants' health care utilization was assessed through a combination of medical record reviews and novel and adapted measures from the Behavioral Risk Factor Surveillance System (BRFSS). Survey self-report data were compared to services and procedures indicated on medical record review.
Time Frame: 6 weeks post-disclosure (approx. 43 weeks after baseline)
Population: 69 participants completed follow-up survey and several participants selected more than one answer for 83 total responses.
Measure: Number; unit: participants
Arm/Group | Healthy Active-Duty Airmen Cohort
Number analyzed (Participants) | 83
participants
  Change in diet | 9
  Change in exercise | 7
  Change in use of vitamin supplements | 5
  Change in use of medication | 5
  Other change | 1
  No change | 56

4. Primary Outcome: Military Healthcare Providers' Genomic Literacy
Description: Military healthcare provider-participants' genomic literacy were measured with a 14-item measure adapted from the ClinSeq Study (Kaphingst K.A. et al. 2012) administered at baseline, before (pre) and immediately after (post) an education session, and at Follow-up near the end of the study. Items are marked as correct (1) or incorrect (0) and summed for a total scale range of 0 to 14, with higher scores indicating higher genomic literacy.
Time Frame: Baseline (pre and post) and Follow-up (follow-up administered approx. 53 weeks after baseline)
Population: Healthcare providers who completed the pre, post and follow-up surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Provider Cohort
Number analyzed (Participants) | 12
score on a scale
  Pre test | 9.92 (1.38)
  Post test | 11.50 (1.45)
  Follow-up | 10.75 (2.25)

5. Secondary Outcome: Active-duty Airmen Attitudes and Perceived Utility Toward Genomic Sequencing
Description: Adapted measures assessed participants' attitudes toward genetic information, trust of physicians and the military regarding use of genetic information. (Hall et al. 2006). Scores are summed, with higher scores on a 4-20 scale representing greater trust.
  A novel survey item at baseline and 6-weeks post-disclosure asked participants to rate the usefulness of whole genome sequencing results for managing health now on a 1-10 scale.
Time Frame: Baseline and 6-weeks post-disclosure (approx.. 43 weeks after baseline)
Population: 69 surveys completed at follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Active-Duty Airmen Cohort
Number analyzed (Participants) | 75
score on a scale
  Trust at baseline | 14.31 (2.47)
  Trust at follow-up | 14.10 (2.25)
  Usefulness - Baseline | 7.76 (2.11)
  Usefulness - follow-up | 7.30 (2.11)

6. Secondary Outcome: Active-duty Airmen's Health Perceptions
Description: Assessed using a validated measure of subjective perceptions about health status. (Latham 2013, DeSalvo 2006). Responses are on a 1 - 5 scale, where higher scores indicate more positive responses.
Time Frame: Baseline and 6-weeks post-disclosure (approx.. 43 weeks after baseline)
Population: 69 surveys were completed at follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Active-Duty Airmen Cohort
Number analyzed (Participants) | 75
score on a scale
  Health perceptions- baseline | 3.95 (0.81)
  Health perceptions - follow-up | 3.86 (0.76)

7. Secondary Outcome: Military Healthcare Providers' Confidence With Genomic Data
Description: Assessed through a scale developed for the Multiplex initiative to measure provider genomic confidence (Gray SW et al 2014). Scores are summed with higher scores on a 5-20 scale indicating greater confidence in military healthcare provider-participants' abilities to understand genetic information
Time Frame: Baseline (pre and post) and Follow-up (follow-up administered approx. 53 weeks after baseline)
Population: Healthcare providers who completed the pre, post and follow-up surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Provider Cohort
Number analyzed (Participants) | 12
score on a scale
  Pre-Test | 7.25 (2.05)
  Post-Test | 13.00 (1.41)
  Follow-up | 12.33 (2.29)

ADVERSE EVENTS:
Time Frame: From baseline survey to approximately 6 weeks after disclosure (43 weeks after baseline)
Description: Any serious adverse events linked to the disclosure of genomic information will be reported both to the Institutional Review Board (IRB) within one week of the time the event is identified. For all other metrics, the PI will review data & report annually to the IRB.
Arm/Group | Healthy Active-Duty Airmen Cohort | Healthcare Provider Cohort
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/12
Other Adverse Events (participants affected / at risk) | 0/75 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03276637/Prot_SAP_000.pdf